CLINICAL TRIAL: NCT06137560
Title: Spectacle Films Utilising S.T.O.P.® Technology for Slowing Down Myopia Progression in Children: A Prospective, Masked, Controlled, Randomised, Clinical Trial.
Brief Title: Spectacle Films Utilising S.T.O.P.® Technology for Slowing Down Myopia Progression in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: nthalmic Pty Ltd (Network)
Collaborators: Zhong Jing Wei Shi (Suzhou) Optical Technology Ltd. (Unknown)
Responsible Party: Principal Investigator, Daniel Tilia, MOptom, PhD, Principal Research Optometrist, nthalmic Pty Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: nthal2021-04
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Assigned Intervention 1 (Active Comparator): Single vision spectacle lens
  Interventions: Device: Single vision spectacle lens
- Assigned Intervention 2 (Experimental): Single vision spectacle lens + S.T.O.P.® Kit 1
  Interventions: Device: Single vision spectacle lens + S.T.O.P.® Kit 1
- Assigned Intervention 3 (Experimental): Single vision spectacle lens + S.T.O.P.® Kit 2
  Interventions: Device: Single vision spectacle lens + S.T.O.P.® Kit 2
- Assigned Intervention 4 (Active Comparator): Static optical signal: single vision spectacle lens + S.T.O.P.® spectacle film
  Interventions: Device: Single vision spectacle lens + S.T.O.P.® Film
- Assigned Intervention 5 (Experimental): Dynamic optical signal: single vision spectacle lens + S.T.O.P.® Kit 1 or 2
  Interventions: Device: Standard single vision spectacle lens + S.T.O.P.® Kit 1 or 2

INTERVENTIONS:
Device: Single vision spectacle lens — Standard single vision spectacle lens
  Arms: Assigned Intervention 1
Device: Single vision spectacle lens + S.T.O.P.® Kit 1 — Standard single vision spectacle lens + S.T.O.P.® Kit 1
  Arms: Assigned Intervention 2
Device: Single vision spectacle lens + S.T.O.P.® Kit 2 — Standard single vision spectacle lens + S.T.O.P.® Kit 2
  Arms: Assigned Intervention 3
Device: Single vision spectacle lens + S.T.O.P.® Film — Standard single vision spectacle lens + S.T.O.P.® Film
  Arms: Assigned Intervention 4
Device: Standard single vision spectacle lens + S.T.O.P.® Kit 1 or 2 — Standard single vision spectacle lens + S.T.O.P.® Kit 1 or 2
  Arms: Assigned Intervention 5

SUMMARY:
There are two parts to this trial. First, to compare the rate of myopia progression of spectacle films using Spatio Temporal Optic Phase (S.T.O.P.®) technology that provide a dynamic optical cue against single vision spectacle lenses. Second, to compare the rate of myopia progression of spectacle films using S.T.O.P.® technology that provide a dynamic optical cue against spectacle films using S.T.O.P.® technology that provide a static optical cue. A dynamic optical cue is one that changes, and a static optical cue is one that does not change.

DETAILED DESCRIPTION:
In the first part of the trial, myopic children (6-14 years of age) will be randomly allocated to wear one of three spectacle lens options (standard single vision spectacle lenses, standard single vision spectacle lenses + S.T.O.P.® Kit 1 spectacle films, or standard single vision spectacle lenses + S.T.O.P.® Kit 2 spectacle films). S.T.O.P.® spectacle films are applied to the front surface of standard single vision spectacle lenses. Both S.T.O.P.® Kits 1 and 2 are comprised of two different sets of spectacle films applied to two different pairs of single vision spectacle lenses which are worn on alternate weeks, and thus both S.T.O.P.® Kits 1 and 2 provide a dynamic optical cue.

In the second part of this trial, participants will be randomly allocated wear of of two spectacle lens options (the best performer from S.T.O.P.® Kits 1 and 2 in terms of reducing the rate of myopic progression and single vision spectacle lenses + S.T.O.P.® film). As previously stated, both S.T.O.P.® Kits 1 and 2 provide a dynamic optical cue while S.T.O.P.® film provide a static optical cue.

The overall trial duration, including follow-up period, is expected to be approximately 42 months. Each participant's duration is expected to be approximately 30 months.

The visits are Baseline, Dispensing, 1 month, 4 months, 6 months, then visits every 6 months after.

All procedures performed at these visits are standard, non invasive clinical tests.

ELIGIBILITY:
Inclusion Criteria:

* Be between 6-14 years inclusive at time of enrolment.
* Have:

  * Read the Informed Assent.
  * Been explained the Informed Assent.
  * Indicated an understanding of the Informed Assent.
  * Signed the Informed Assent.
* Have their parent / legal guardian:

  * Read the Informed Consent.
  * Been explained the Informed Consent.
  * Indicated an understanding of the Informed Consent.
  * Signed the Informed Consent.
* Along with their parent / legal guardian, be capable of comprehending the nature of the study, and be willing and able to adhere to study requirements.
* Along with their parent / legal guardian, agree to maintain the visit and prescribed wearing schedule.
* Agree to wear allocated spectacles for a minimum of 5 days per week, at least 6 hours per day for the duration of the study and to inform the investigator if their schedule is interrupted.
* Possess wearable and visually functioning spectacles.
* Be in good general health, based on the parent's / legal guardian's knowledge.
* Have best-corrected high contrast visual acuity based on manifest refraction of 0.10 logMAR (20/25, 6/7.6) or better in each eye.
* Meet the following criteria determined by cycloplegic autorefraction at Baseline:

  * -5.00 D ≤ spherical equivalent ≤ -0.75 D and sphere component ≤ -0.50 DS.
  * -1.50 DC ≤ astigmatic component ≤ 0 DC.
  * |Spherical equivalent anisometropia| ≤ 1.00 D.

Exclusion Criteria:

* Participant is currently, or within 30 days prior to this study, has been an active participant in another study.
* Current or prior use of ANY form of myopia control, including but not limited to:

  * Optical devices:

    * Bifocal or multifocal spectacles of any type.
    * Bifocal or multifocal contact lenses of any type.
    * Orthokeratology of any type.
  * Pharmacological agents:

    * Atropine with a concentration > 0.01%. Participants who have previously used 0.01% atropine are eligible for this study provided they agree not to use 0.01% atropine for at least 30 days before baseline and at any time during the study.
    * Pirenzepine
* Participant born earlier than 30 weeks or weighed < 1500 g at birth.

  * A verbal report from the participant's parent / legal guardian is sufficient.
* Habitual use of a systemic or topical medication that may alter normal ocular findings / is known to affect a participant's ocular health / physiology either in an adverse or beneficial manner at enrolment and / or during the clinical trial.
* A known allergy to sodium fluorescein, benoxinate, proparacaine, tropicamide, or cyclopentolate.
* Strabismus as determined by cover test at distance (≥ 3 m) or near (40 cm) while wearing distance correction under non-cycloplegic conditions.
* Known ocular or systemic disease, such as but not limited to:

  * Diabetes.
  * Graves' disease.
  * Glaucoma.
  * Uveitis.
  * Scleritis.
  * Auto immune diseases such as ankylosing spondylitis, multiple sclerosis, Sjogrens syndrome, and systemic lupus erythematosus.
* Any ocular, systemic, or neuro-developmental conditions that could influence refractive development, such as but not limited to:

  * Persistent pupillary membrane.
  * Vitreous haemorrhage.
  * Cataract.
  * Central corneal scarring.
  * Eyelid haemangiomas.
  * Marfan's syndrome.
  * Down's syndrome.
  * Ehler's-Danlos syndrome.
  * Stickler's syndrome.
  * Ocular albinism.
  * Retinopathy of prematurity.
* Keratoconus or irregular cornea.
* The investigator may, at their discretion, exclude anyone who they believe may not be able to fulfil the clinical trial requirements or it is believed to be in the participant's best interests.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Axial length | Baseline, First Dispense (up to 26 days from Baseline), then 1 month, 4 months, and 6 months after First Dispense
  Difference in change from Baseline in axial length between single vision (control) and S.T.O.P.® Kit 1 & 2 (tests)
Axial length | Second Dispense (up to 392 days from Baseline), then 6 months, 12 months, and 18 months after Second Dispense
  Difference in change from Second Dispense in axial length between static optical cue (control) and dynamic optical cue (test)

SECONDARY OUTCOMES:
Cycloplegic spherical equivalent autorefraction | Baseline, First Dispense (up to 26 days from Baseline), then 1 month, 4 months, and 6 months after First Dispense
  Difference in change from Baseline in cycloplegic spherical equivalent autorefraction between single vision (control) and S.T.O.P.® Kit 1 & 2 (tests)
Cycloplegic spherical equivalent autorefraction | Second Dispense (up to 392 days from Baseline), then 6 months, 12 months, and 18 months after Second Dispense
  Difference in change from Second Dispense in cycloplegic spherical equivalent autorefraction between static optical cue (control) and dynamic optical cue (test)
Visual performance as measured by high contrast visual acuity at 6 m | 1 month, 4 months, and 6 months after First Dispense (up to 26 days from Baseline)
  Difference in visual performance between single vision (control) and S.T.O.P.® Kit 1 & 2 (tests)
Visual performance as measured by high contrast visual acuity at 6 m | 6 months, 12 months, and 18 months after Second Dispense (up to 392 days from Baseline)
  Difference in visual performance between static optical cue (control) and dynamic optical cue (test)
Visual performance as measured by a non validated questionnaire based on a 1-10 | 1 month, 4 months, and 6 months after First Dispense (up to 26 days from Baseline)
  Difference in visual performance between single vision (control) and S.T.O.P.® Kit 1 & 2 (tests)
Visual performance as measured by a non validated questionnaire based on a 1-10 | 6 months, 12 months, and 18 months after Second Dispense (up to 26 days from Baseline)
  Difference in visual performance between static optical cue (control) and dynamic optical cue (test)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Tilia, Optom, PhD, Principal Investigator — nthalmic Pty Ltd
Locations (5):
- China (2):
  - Tianjin Eye Hospital, Tianjin, Heping District
  - Shanghai Fudan University Eye and ENT Hospital, Shanghai, Xuhui District
- India (3):
  - Divyajyoti Trust Tejas Eye Hospital, Surat, Gujarat
  - LV Prasad Eye Institute, Hyderabad, Telangana
  - Pristine Eye Hospitals, Hyderabad, Telangana

IPD SHARING:
Plan to Share IPD: No